CLINICAL TRIAL: NCT01019837
Title: Efficacy and Safety of Vaccination Against Influenza H1N1 in Patients With Inflammatory Bowel Diseases Treated With Immunomodulators and Biologics
Brief Title: Efficacy and Safety of Vaccination Against Influenza H1N1 in Patients With Inflammatory Bowel Diseases (IBD) Treated Immunomodulators and Biologics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-09-ID-553-CTIL
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Influenza H1N1
Keywords: Vaccine
MeSH Terms: interventions — focetria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Monovalent MF59- Adjuvanted vaccine (Experimental): Focetria (Monovalent MF59-Adjuvanted vaccine) 7.5 mcg Hemagglutinin H1/InfluezaA/California/7/2009 ,9.75 mg squalene MF59, 1.175 mg polysort80, 1.175 mg sorbitan trioleate Intra muscular
  Interventions: Biological: Focetria (Monovalent MF59-Adjuvanted vaccine)

INTERVENTIONS:
Biological: Focetria (Monovalent MF59-Adjuvanted vaccine) — Biological: Focetria (Monovalent MF59-Adjuvanted vaccine)

SUMMARY:
The spread of Influenza H1N1 has prompted the development of vaccines against this virus. IBD patients are at increased risk of developing complications of Influenza H1N1. The efficacy and safety of H1N1 vaccination have not been evaluated in this population of patients. We would like to estimate the efficacy and safety of vaccination against influenza H1N1 in patients with IBD who treated with immunomodulatory drugs.

DETAILED DESCRIPTION:
200 patients with IBD and 200 healthy subjects will participate in the study. All the subjects will be vaccinated with Focetria (Novartis) and will be evaluated the day of vaccination and 4 weeks later.

The evaluation will include:

Efficacy of the vaccine: Blood will be drawn on day 0 and 4 weeks later and tested for the presence of antibodies against A/California17/2009/H1N1 by hemagglutination inhibition test.

Safety of the vaccine:

* Records of adverse event
* Assessment of disease activity : CDAI and MAYO score

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from IBD (inflammatory bowel disease): UC/ CD
2. Able to firm an informed consent
3. Aged - 18-65
4. Candidates to receive vaccination against H1N1, according to the recommendation of the Ministry of Health
5. patients who treated with immunomodulators and biologics

Exclusion Criteria:

1. Allergy to eggs
2. Known allergy to seasonal influenza vaccine
3. Pregnant women
4. Patients who inoculate another vaccine in the past 3 weeks (except vaccine fot seasonal influenza
5. Patients without worsening in their disease condition (stable condition)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who will achieve a titer of antibodies above 1/40 within the groups of patients in comparison with healthy subjects | 4 weeks

SECONDARY OUTCOMES:
Safety of the vaccine with regard to disease activity by changes in Crohn's Disease Activity Index (CDAI) and MAYO score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iris Dotan, Dr., Study Director — Tel-Aviv Sourasky Medical Center